CLINICAL TRIAL: NCT04564534
Title: Impact of Pre-procedure Cognitive Status on Outcome at 3 Months After Transcatheter Aortic Valve Implantation
Acronym: TAVI-Geriatrie
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2019/417
Record Dates: First submitted 2019-06-20; First posted 2020-09-25 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Aortic Stenosis
Keywords: transcatheter aortic valve replacement; aortic stenosis; cognitive status
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be taken and centrifuged, and plasma will be aliquoted and frozen at -80°Celsius for analysis of growth differentiation factor (GDF) 15.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study cohort: Adult (>18 years) patients with aortic stenosis in whom TAVI is planned and who perform their pre-TAVI work-up in our centre will be invited to undergo cognitive assessment using the MoCA at the time of their hospitalization for pre-TAVI work-up.
  The MoCA will be administered by trained professionals with MoCA certification.
  Clinical outcomes, as assessed by the VARC2 criteria, will be collected for all patients at 3 months after the TAVI procedure.
  Interventions: Other: MoCA cognitive assessment

INTERVENTIONS:
Other: MoCA cognitive assessment — cognitive assessment using the validated MoCA test administered via an application on an iPad

SUMMARY:
This study plans to investigate the relationship between cognitive status pre-procedure, and clinical outcomes at 3 months in patients undergoing transcatheter aortic valve implantation (TAVI).

DETAILED DESCRIPTION:
This study plans to investigate the relationship between cognitive status pre-procedure, as assessed using the Montreal Cognitive Assessment (MoCA) administered on a tablet, and clinical outcomes at 3 months as assessed by the VARC2 criteria, in patients undergoing transcatheter aortic valve implantation (TAVI)

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over
* Scheduled to undergo TAVI
* Provide informed consent
* Able to understand French

Exclusion Criteria:

* subjects under legal guardianship or other legal protection
* subjects with documented severe dementia
* subjects with anticipated poor compliance
* subjects unable to understand French sufficiently well to perform the MoCA test
* pregnant women
* subjects within the exclusion period of another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with aortic stenosis and a confirmed indication for TAVI, scheduled to undergo TAVI and who perform their pre-TAVI work-up in our centre will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
All-cause death | through 30 days after the TAVI procedure
  Safety outcome at 3 months as assessed by the VARC2 criteria: all-cause death
Stroke | through 30 days after the TAVI procedure
  Safety outcome at 30 days as assessed by the VARC2 criteria: stroke
life-threatening bleed | through 30 days after the TAVI procedure
  Safety outcome at 30 days as assessed by the VARC2 criteria: life-threatening bleed
Combined VARC2 safety outcome | through 30 days after the TAVI procedure
  Safety criteria (within 30 days of the procedure) include all-cause death; stroke; life-threatening bleed; renal insufficiency; coronary artery obstruction requiring intervention; major vascular complication; valve dysfunction.
  Clinical Efficacy criteria (30 days to 3 months after the procedure) include: all-cause death; stroke; re-admission for valve-rela
Combined VARC2 efficacy outcome | through 30 days after the TAVI procedure
  Clinical Efficacy criteria (30 days to 3 months after the procedure) include: all-cause death; stroke; re-admission for valve-related symptoms or worsening heart failure; NYHA Class III or IV; valve-related dysfunction.

SECONDARY OUTCOMES:
Time required for MoCA | At the time of MoCA completion
  Length of time required to administer the MoCA test using a tablet
Biological parameters pre-procedure | pre-procedure
  Blood count; prothrombin; TCA; fibrinogen; INR; creatinine; CRP; BNP; TSH; HbA1c; troponin; albumin; GDF15.
Relationship between MoCA score and each component of the VARC2 | At 3 months after TAVI procedure
  The relationship between the MoCA and each individual component of the VARC2 will be investigated in bivariable analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Francois Schiele, MD, PhD, Principal Investigator — CHRU Besancon
Locations (1):
- University Hospital Jean Minjoz, Besançon, France

IPD SHARING:
Plan to Share IPD: No